CLINICAL TRIAL: NCT01917487
Title: A Trial to Evaluate the Precision and Accuracy of the NBM-200 Series When Used in a Continuous Prospective Mode
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: OrSense, Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: QD04.5.1-25
Record Dates: First submitted 2013-08-01; First posted 2013-08-06 (Estimated); Last update posted 2013-09-10 (Estimated); Status verified 2013-09

CONDITIONS: Anemia
MeSH Terms: conditions — Anemia

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of the study is to define the precision, accuracy and variability of the NBM-200 system in non invasive blood Hemoglobin (Hb) measurements relative to the laboratory blood analyzer by comparing two consecutive Hb values obtained by the NBM system to venous values.

DETAILED DESCRIPTION:
Each subject will be placed in a comfortable position in a temperature regulated room. Participants will have two consecutive non invasive (NBM) measurements taken which involves inserting the thumb into a ring shaped sensor. After each non invasive measurement the sensor will be removed. Each measurement takes approximately 85 seconds and involves the finger cuff inflating (to over systolic pressure) and deflating several times in quick successions in order to measure and calculate the Hb values. The two non invasive measurements will be performed using the same finger. After the NBM system testing is complete and recorded, the subject will have a venous (venipuncture) blood sample collected in order to provide two blood tests performed on two different models of routine automated complete blood count or Hb blood analyzers.

Addendum:

Reproducibility Procedure (optional) Each subject will be measured by each one of the three operators, three NBM system units, 3 times consecutively (without removal) on his right thumb and right index finger. The order of each measurement sequence will be randomized (thumb/index). There will be an intermission of 3 to 5 minutes between the 3 measurement sets taken on each participant. In case of a longer intermission, the subject will be measured again and the previous results will be excluded.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years and over
* Healthy volunteers
* Anemia patients

Exclusion Criteria:

* Participants under the age of 18 years
* Patients with significant deformity, degenerative changes or oedema of the thumb or index fingers
* Patients with localized infection, ulceration or skin breaks involving the fingers
* Patients with vascular disease or Raynaud's phenomenon affecting the fingers
* Participants who are unable to give informed written consent
* Pregnancy

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: healthy volunteers and oncology patients
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2011-11; Primary Completion 2013-10 (Estimated); Study Completion 2013-11 (Estimated)

PRIMARY OUTCOMES:
Compare the Hb values from the Noninvasive Blood Monitor(NBM200) series against the Hb from the lab blood analyser on healthy volunteers and oncology patients | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Ohad Cohen, Prof., Principal Investigator — The Chaim Sheba Medical Center at Tel Hashomer
Locations (1):
- The Chaim Sheba Medical Center at Tel Hashomer, Ramat Gan, Israel, Israel